CLINICAL TRIAL: NCT03482596
Title: The Effects of Reducing Prolonged Sitting Bouts With Regular Light Upright Movement Breaks on Glucose Regulation in Individuals at High Risk of or With Type 2 Diabetes
Brief Title: The Effects of Reducing Prolonged Sitting Bouts in Individuals at High Risk of or With Type 2 Diabetes
Acronym: UP FOR 5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other); Loughborough University (Other); Baker Heart and Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0641
Record Dates: First submitted 2018-03-05; First posted 2018-03-29 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Sedentary Behaviour; Prevention
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All participants will follow the personalised multifaceted intervention to reducing/breaking prolonged sitting.
  Interventions: Behavioral: Reducing/breaking prolonged sitting

INTERVENTIONS:
Behavioral: Reducing/breaking prolonged sitting — The participants will be encouraged to reduce prolonged sitting by at least 60 minutes per day by introducing light upright movement breaks spread throughout their day. The frequency and duration of these breaks will be tailored to each participant to suit their individual circumstances.
  The intervention will involve education regarding the health implications of prolonged sitting, personalised goal setting, behavioural feedback and self-monitoring of behaviour.

SUMMARY:
Over 3 million in the United Kingdom are now diagnosed with type 2 diabetes, with current estimates suggesting this will rise to over 5 million by 2025. Type 2 diabetes increases the risk of developing cardiovascular disease, kidney disease, depression, neuropathy and dementia, along with being a leading cause of amputation and adult blindness.

Sedentary behaviour, defined as any waking moment spend sitting or reclining with energy expenditure equal to or less than 1.5 METs, has emerged as a risk factor in the development of type 2 diabetes. Recent evidence has shown that breaking up prolonged sitting with regular short bouts of activity or standing lower postprandial glucose and insulin. However, the effectiveness of breaking prolonged sitting on glucose metabolism over a longer period of time is unknown. Therefore, the aim of this study is to investigate whether the reduction in postprandial plasma glucose in response to breaking prolonged sitting time is maintained following an intervention to reduce and break up prolonged sitting over a four to five week period.

The study will be a single group intervention with pre and post randomised measurement conditions (prolonged sitting and light upright breaks) at both time points. A sample of 43 people (34 to complete), aged 50-75, identified as at risk of or with (drug naive) type 2 diabetes will be sought. The intervention will last approximately 5 weeks. Experimental conditions will be conducted before and after the intervention to assess whether reducing and breaking up prolonged sitting in free living effects glucose metabolism.

DETAILED DESCRIPTION:
Study Design

This study consists of an intervention lasting approximately 5 weeks (depending on follow-up measurement timings), with a before and after 'two-arm' randomised crossover design, one prior to the intervention and one at the end of the intervention used as measurement periods. Screening will require one laboratory visit, with the study commencing one week following baseline. The intervention will last a minimum of four weeks, while the measurement conditions will each involve two laboratory days separated by a minimum of five days. The duration from screening through to study end will be an estimated 9 weeks. This trial will evaluate the effectiveness of regular light upright movement breaks at reducing glucose iAUC by examining if acute adaptations to sitting time are maintained or improved following the behavioural intervention.

Study Setting

The study will be co-ordinated within the Leicester Biomedical Research Centre (Leicester Diabetes Centre) at the Leicester General Hospital. Clinical measurement sessions will be carried out by the appointed research team. Participants will be asked to visit the study centre on seven occasions.

Measurement conditions

Measurement condition A will consist of seven and a half hours of prolonged sitting, where participants will be restricted from walking or standing for the duration. Lavatory breaks will be carried out using a wheelchair to transport the participant to minimise time spent upright. The condition will be conducted in the laboratory at the Leicester Diabetes Centre. Participants will have access to a computer with internet services, books and magazines for the duration of the measurement day.

Upon arrival, the participant will have a cannula inserted into an accessible vein by a trained member of the study team, which will be used to collect blood samples throughout the measurement day. Blood pressure will be taken prior to each blood sample, while visual analogue scales for hunger, energy, fullness, satiety, desire to eat and fatigue will be completed following each blood sample. The first blood sample will be taken at the start of the 'steady state' following anthropometric measurements. The next sample will be taken one hour after the first sample. Following this, participants will be given a standardized meal consumed over a maximum of 15 minutes. Blood samples will be then be taken at 30, 60, 120 and 180 minutes after commencing eating. Another standardized meal and the same schedule of blood sampling will take place following the blood sample taken 180 minutes postprandial to the first meal. Meals will be based on body weight, with eight kcals per kg of body weight, made up of 52% carbohydrate, 35% fats and 13% protein.

Measurement condition B will follow the same procedures as condition A in terms of standardised meals, blood sampling, blood pressure, visual analogue scales and meal consumption. Similarly, participants will be allowed access to a lavatory in the same way as condition A, as well as have access to a computer, books, magazines and other typical sedentary pursuits. The only difference in this measurement condition to condition A, is that participants will regularly break their sitting time, for five minutes every 30 minutes with upright light movement after sitting quietly for one hour upon arrival and following cannulation (steady state). This will involve the participant walking and moving around slowly and freely in the testing room and surrounding laboratory. This is to maximise the ecological validity of the study, particularly in comparison to studies using a treadmill for light walking breaks. Five minute breaks every 30 minutes was chosen as this has previously shown positive effects on both glucose metabolism and insulin in postmenopausal women (19). Light breaks will accumulate 60 minutes of light upright movement across the measurement day.

Intervention

The participants will be encouraged to reduce prolonged sitting by at least 60 minutes per day by introducing light upright movement breaks spread throughout their day. The frequency and duration of these breaks will be tailored to each participant to suit their individual circumstances. A 60 minute reduction is judged to be clinically meaningful. For example, a modelling study found that replacing 60 minutes of sedentary time with light movement was associated with around 20% better insulin sensitivity in those with dysglycemia.

The intervention will involve one participant face-to-face session, lasting approximately two hours. It will also involve personalised feedback which will review progress and goals based on the baseline data. The visit will involve personalised education and goal setting, based on objective measures of sitting time taken at baseline. These data will be explained to the participant, which will then form the basis of a plan to reduce prolonged bouts of sitting with light movement. This session will also explain what is meant by light movement, as well as identifying a number of different ways to break prolonged bouts effectively. Participants will be encouraged to self-monitor their sitting time, with specific examples of how his can be achieved depending on the needs of the participant. They will be given an accelerometer to be worn for the duration of the four week intervention.

The participant will receive feedback from a member of the study team on at least a weekly basis (more frequently feedback expected in the early weeks) in regards to current sedentary behavior and movement time. Data received from the accelerometer or self-monitoring device will be used to discuss the positives and negatives of the previous days or week's behaviour. These will be talked through and adjustments made to the goals if needed. The feedback sessions will take place primarily over the telephone, however if the participant would like to visit the Leicester Diabetes Centre for these sessions that will be made available to them. All feedback is personalised meaning it will be different for each participant in terms of the data fed back as well as the timings of each feedback session

ELIGIBILITY:
Inclusion Criteria:

* Male and Postmenopausal Females.
* ≥ 40 to ≤ 75 years of age.
* And either:

  * Overweight (White: BMI > 25 - <30, South Asian, Black or Chinese: > 23 <27.5) with HbA1c between 6.0 and 7.5%, within the previous 36 months).
  * Obese (White: BMI ≥ 30, South Asian, Black or Chinese: ≥ 27.5).
* Large proportions of their day spent sitting (self-reported).
* Participant is willing and able to give informed consent to take part in the study.
* Not planning on altering their diet during the study.
* Able to walk without the use of an assistive device or requiring assistance form another person

Exclusion Criteria:

* The participant may not enter the study if ANY of the following apply:
* Reporting taking part in regular (at least once a week) sport of strenuous exercise.
* HbA1c > 7.5%.
* Overweight with HbA1c < 6.0%.
* Taking any glucose lowering therapies.
* Type 1 diabetes.
* Recent cardiovascular event (within the last 12 months).
* Female premenopausal.
* Current smoker.
* Terminal illness.
* Steroid use.
* Comorbidity that the research team consider to be a contraindication to involvement in the study
* Unable to communicate in English.
* Unable to provide written informed consent.

In the circumstance that an individual is not sure whether they meet the inclusion/ exclusion criteria, they will be reviewed by a named medic on the delegation of authority log for a clinical decision to be made during the baseline visit.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females may only be eligible if they are postmenopausal
Enrollment: 43 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
Glucose incremental Area Under the Curve (iAUC) | Assessed via 10 blood samples.Two of which will be taken while fasting and the remainder taken at 30, 60, 120 and 180 minutes following both breakfast and lunch meals. This will be assessed for all of the 7.5 hour experimental treatment conditions
  Glucose iAUC will be used to assess whether, following the intervention, the expected improvement in glucose metabolism is maintained or improved in the post-measurement conditions compared to the pre-measurement conditions.

SECONDARY OUTCOMES:
Insulin incremental Area Under the Curve (iAUC) | Assessed via 10 blood samples.Two of which will be taken while fasting and the remainder taken at 30, 60, 120 and 180 minutes following both breakfast and lunch meals. This will be assessed for all of the 7.5 hour experimental treatment conditions
  iAUC will be used to assess whether, following the intervention, the expected reduction in insulin is maintained or improved in the post-measurement conditions compared to the pre-measurement conditions.
Triglycerides incremental Area Under the Curve (iAUC) | Assessed via 10 blood samples.Two of which will be taken while fasting and the remainder taken at 30, 60, 120 and 180 minutes following both breakfast and lunch meals. This will be assessed for all of the 7.5 hour experimental treatment conditions
  iAUC will be used to assess whether, following the intervention, the expected reduction in triglycerides is maintained or improved in the post-measurement conditions compared to the pre-measurement conditions.
Blood pressure incremental Area Under the Curve (iAUC) | Assessed prior to all 10 blood samples. This will be assessed for all of the 7.5 hour experimental treatment conditions
Acylated ghrelin | Assessed via 5 blood samples, One of which is taken fasted and the remainder taken at 30, 60, 120 and 180 minutes following breakfast during condition A
  Appetite hormone
Total PYY | Assessed via 5 blood samples, One of which is taken fasted and the remainder taken at 30, 60, 120 and 180 minutes following breakfast during condition A
  Appetite hormone
Subjective appetite - Hunger | Assessed after each blood sample during every experimental condition. Through study completion, an average of 9 weeks.
  Measure via a visual analog scale. Scale ranges from 0 to 100. The higher the number the more hungry the person feels.
Subjective appetite - Fullness | Assessed after each blood sample during every experimental condition. Through study completion, an average of 9 weeks.
  Measure via a visual analog scale. Scale ranges from 0 to 100. The higher the score, the more full a person feels.
Subjective appetite - Satiety | Assessed after each blood sample during every experimental condition. Through study completion, an average of 9 weeks.
  Measure via a visual analog scale. Scale ranges from 0 to 100. The higher the score, the more satisfied a person feels.
Subjective appetite - Quantity | Assessed after each blood sample during every experimental condition. Through study completion, an average of 9 weeks.
  Measure via a visual analog scale. Scale ranges from 0 to 100. The higher the score, the more someone believes they can eat.
Fatigue (acute) | Assessed after each blood sample during every experimental condition. Through study completion, an average of 9 weeks.
  Measure via a visual analog scale, one for energy and one for fatigue. Scale ranges from 0 to 100. The higher the number, the more fatigued someone feels.
Energy (acute) | Assessed after each blood sample during every experimental condition. Through study completion, an average of 9 weeks.
  Measure via a visual analog scale, one for energy and one for fatigue. Scale ranges from 0 to 100. The higher the number, the more energetic someone feels
Fasting glucose | Before and after the intervention. Through study completion, an average of 9 weeks.
Fasting insulin | Before and after the intervention. Through study completion, an average of 9 weeks.
Fasting triglycerides | Before and after the intervention. Through study completion, an average of 9 weeks.
Fasting IL-6 | Before and after the intervention. Through study completion, an average of 9 weeks.
Cholesterol | Before and after the intervention. Through study completion, an average of 9 weeks.
HDL Cholesterol | Before and after the intervention. Through study completion, an average of 9 weeks.
LDL Cholesterol | Before and after the intervention. Through study completion, an average of 9 weeks.
Fasting creatinine | Before and after the intervention. Through study completion, an average of 9 weeks.
  Serum creatinine is an important indicator of renal health because it is an easily measured by-product of muscle metabolism that is excreted unchanged by the kidneys.
Mood | Baseline and last week of the intervention. Through study completion, an average of 9 weeks.
  Profile of Mood States
Depressive symptoms | Baseline and last week of the intervention. Through study completion, an average of 9 weeks.
  Center for Epidemiologic Studies Depression Scale
Chronic fatigue | Baseline and last week of the intervention. Through study completion, an average of 9 weeks.
  Chalder Fatigue Scale
Average blood glucose | Week following baseline and during the last week of the intervention. Through study completion, an average of 9 weeks.
  Measure via continuous glucose monitors
Time spent in hypoglycemia | Week following baseline and during the last week of the intervention. Through study completion, an average of 9 weeks.
  Measure via continuous glucose monitors
Time spent in hyperglycemia | Week following baseline and during the last week of the intervention. Through study completion, an average of 9 weeks.
  Measure via continuous glucose monitors
Physical function | Baseline and at the end of the intervention. Through study completion, an average of 9 weeks.
  Measure via a battery of tests: The MINIBESTest, 30 second chair sit stand test, 20 meter walk test and grip strength.
Adherence to the intervention | Data during the intervention period will be compared to baseline. Through study completion, an average of 9 weeks.
  Measure via accelerometer
Physical behaviours | Data during the intervention period will be compared to baseline. Through study completion, an average of 9 weeks.
  sleep, sitting, standing, stepping
Sedentary time | Data during the intervention period will be compared to baseline. Through study completion, an average of 9 weeks.
  Accelerometer sedentary time
Light intensity physical activity | Data during the intervention period will be compared to baseline. Through study completion, an average of 9 weeks.
  Accelerometer derived Light intensity physical activity
Moderate to vigorous intensity physical activity (MVPA) | Data during the intervention period will be compared to baseline. Through study completion, an average of 9 weeks.
  Accelerometer derived moderate intensity activity and vigorous intensity activity. These will be combined to created one variable, MVPA
Sleep | Data during the intervention period will be compared to baseline. Through study completion, an average of 9 weeks.
  Sleep will be derived from the accelerometer wear diaries.
Intervention perception | Conducted at the end of the intervention. Through study completion, an average of 9 weeks.
  Interviews

CONTACTS AND LOCATIONS:
Locations (1):
- Leicester Diabetes Centre, Leicester, Leicestershire, United Kingdom